CLINICAL TRIAL: NCT05491343
Title: Management of Uterine Arteriovenous Malformation- a Comparison of 2 Management Possibilities- Observation vs. Progesterone Treatment/ a Randomized Control Trial
Brief Title: Observation vs Progesterone Treatment for Management of Uterine Arteriovenous Malformation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Etty Spiegel, Dr., HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0060-22EMC
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Arteriovenous Malformations
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Medroxyprogesterone; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Conservative management (No Intervention)
- Progesterone treatment (Experimental)
  Interventions: Drug: MedroxyPROGESTERone Injection [Depo-Provera]; Device: Other

INTERVENTIONS:
Drug: MedroxyPROGESTERone Injection [Depo-Provera] — The drug-induced endometrial changes would likely to prevent the shedding of endometrium, in turn preventing the exposure of AVM.
  Arms: Progesterone treatment
Device: Other — Follow up using US
  Arms: Progesterone treatment

SUMMARY:
A randomized trial which compares conservative management to progesterone based treatment for arteriovenous malformation

ELIGIBILITY:
Inclusion Criteria:

* women between age of 18 to 50, diagnosed with AVM
* hemodynamically stable at clinical presentation

Exclusion Criteria:

* unstable patients
* contraindication to treatment
* US examination not in the US department

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
AVM regression | 3 weeks
  The time from diagnosis to regression

IPD SHARING:
Plan to Share IPD: Yes